CLINICAL TRIAL: NCT04979390
Title: A Phase 1 Study to Evaluate the Safety, Tolerability and Pharmacokinetics of New Formulation SHR-1316 in Subjects With Advanced Tumors
Brief Title: Safety, Tolerability and Pharmacokinetics of the New Formulation SHR-1316 in Subjects With Advanced Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SHR-1316-I-103
Record Dates: First submitted 2021-07-12; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: SHR-1316 administrated intravenously (IV) at protocol defined dose levels
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Drug: SHR-1316

INTERVENTIONS:
Drug: SHR-1316 — SHR-1316 administrated intravenously (IV) at protocol defined dose levels

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of the new formulation SHR-1316 in subjects with advanced tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Histologically or cytologically confirmed advanced cancer in patients who are fail to current standard therapy or lack of effective therapy.
3. Estimated life expectancy ≥12 weeks.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Adequate organ functions.
6. If of childbearing potential (male or female), agrees to practice an effective form of contraception during study treatment and for at least 3 months following last treatment dose.
7. Patients must be willing and able to provide written informed consent prior to the performance of any study-specific procedure.

Exclusion Criteria:

1. Known history of hypersensitivity to any components of the SHR-1316 product.
2. Patient- Prior treatment with the following agents:

   1. "Check-point inhibitors", including Programmed death receptor-1 (PD-1), PD-L1;
   2. Receipt of investigational agents within 4 weeks prior to study treatment;
   3. Current treatment on another therapeutic clinical trial, unless the observational (non-interventional) clinical trials or follow-up of interventional clinical trials;
   4. Any anti-cancer therapy (including chemotherapy, immunotherapy, hormone therapy, target therapy, biotherapy or tumor embolization), administered within 4 weeks prior to study treatment; or within 6 weeks in the case of certain therapies (e.g., mitomycin C and nitrosoureas). Any such, unless discussed and explained with the sponsor;
   5. Anticipated need for any anti-cancer therapy (including chemotherapy, immunotherapy, hormone therapy, or biotherapy) during SHR-1316 treatment; except palliative radiotherapy;
   6. Receipt of any anti-cancer vaccines; receipt of immunomodulatory drugs within 4 weeks prior to study treatment; topical, nasal spray and inhaled corticosteroids as well as systemic steroid therapy in physiological doses (such as: prednisone ≤10 mg/day) are acceptable.
3. Patients have unrecovered (ie, to NCI CTCAE grade ≤1) from all toxicity associated with previous treatments (exception: patients may enter with continuing alopecia irrespective of CTCAE grade; grade 2 peripheral nerve diseases).
4. Known Active central nervous system (CNS) metastases; Patients who had previously received brain or meningeal metastasis therapy, who were clinically stable for at least 8 weeks, and who had stopped systemic sex hormone therapy (such as： prednisone > 10 mg/day) for more than 4 weeks were included.
5. Subjects with active autoimmune disease, history of autoimmune diseases, including but not limited to myasthenia gravis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, etc.
6. Active or history of immune deficiency, such as human immunodeficiency virus (HIV) infection; History of organ transplantation.
7. History or evidence of cardiovascular (CV) risk including any of the following: Congestive heart failure (Class >2) as defined by the New York Heart Association functional classification system (NYHA), unstable angina pectoris, Recent (within the past 12 months) history of myocardial infarction, clinically significant supraventricular or ventricular arrhythmias need treatment or intervention.
8. Patients with clinically significant ECG abnormalities (QT interval corrected for rate by Fridericia's formula [QTcF] >470 msec for female and >450 msec for male on the ECG obtained at Screening).
9. Active infection that need drug intervention or an unexplained fever >38.5°C (fever caused by cancer can be included according to the judgement of the researcher).
10. Active pulmonary tuberculosis infection.
11. Positive for Hepatitis B or C.
12. Known history of psychoactive drug abuse, alcohol abuse or drug use.
13. Known history of any other malignant cancer within past 3 years. Exceptions: completely resected basal cell carcinoma and squamous cell carcinoma of the skin; and completely resected carcinoma in situ of cervix.
14. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-08-10 (Estimated); Primary Completion 2022-02-10 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse events/serious adverse events (based on NCI-CTC AE 5.0) | approximately 1 year
Maximum plasma concentration (Cmax) | approximately 1 year
Time to maximum concentration (Tmax) | approximately 1 year
Area under the concentration-time curve from time zero to time（AUC0-t） | approximately 1 year
Area under the concentration-time curve extrapolated to infinity (AUC0-∞.) | approximately 1 year
Elimination half-life (t1/2) | approximately 1 year
Clearance (CL) | approximately 1 year
Volume of distribution (Vz) | approximately 1 year
Trough concentration (Cmin) | approximately 1 year
Accumulatio of ratio (Rac) | approximately 1 year

SECONDARY OUTCOMES:
Immunogenicity of SHR-1316 | approximately 1 year
  Anti-SHR-1316 antibody (ADA), neutralizing antibody (Nab)
Objective response rate (ORR) | approximately 1 year
Progression-free survival (PFS) | approximately 1 year
Duration of response (DoR) | approximately 1 year
Disease control rate (DCR) | approximately 1 year
Overall survival (OS) | approximately 1 year